CLINICAL TRIAL: NCT02934074
Title: Investigating the Relationship Between Gait Variability and Related Factors in Individuals With Lower Limb Loss
Brief Title: Relationship Between Gait Variability and Sensation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD,PT, Hacettepe University
Other Study IDs: GO 16/344
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Amputation, Traumatic
Keywords: Limb Loss; Gait Variability; Phantom Sensation; Phantom Pain; Peripheral Sensation
MeSH Terms: conditions — Amputation, Traumatic; Phantom Limb

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days

GROUPS / COHORTS (1):
- Unilateral Lower Limb Loss: Individuals with unilateral lower limb loss will be participants of the group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Twenty individuals who were referred to receive physiotherapy will be participants of the study. Participants with lower limb loss will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, year, side and level of limb loss will be recorded. Gait parameters (step length, variation of step length) will evaluate with Gait Trainer Biodex 2, at participant's preferred speed.Phantom sensation and phantom pain will be asked as existence or not. Sensorial loss will evaluate with Semmes Weinstein Monofilaments

DETAILED DESCRIPTION:
Twenty participants with lower limb loss who were referred to receive amputee rehabilitation at Hacettepe University, Faculty of Health Sciences, department of Physiotherapy and Rehabilitation, Prosthetics and Biomechanics unit, will be the subjects of this study.

Participants with lower limb loss will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, year, side and level of limb loss will be recorded. Gait parameters (step length, variation of step length) will evaluate with Gait Trainer Biodex 2, at participant's preferred speed. To eliminate the learning effect, participants practiced at treadmill to determine appropriate gait speed. Once participants implied the preferred speed, they asked to walk at their self selected speed for 6 minutes. Data was recorded between the 2nd and 4th minutes at walk. Phantom sensation and phantom pain will be asked as existence or not. Sensorial loss will evaluate with Semmes Weinstein Monofilaments.

ELIGIBILITY:
Inclusion Criteria:

Individuals with unilateral lower limb loss Traumatic limb loss Age between 20-55 years Using conventional type socket design Dynamic foot using

Exclusion Criteria:

Have passive joint limitation at extremities Surgery at last 1 year Systemic problems such as neurologic disorders, rheumatoid disorders… Another orthopedic anomalies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with traumatic lower limb loss
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Step length variability assesment while walking. | Initially evaluation at first minute
  Gait parameters (step length, variation of step length) will be evaluated with Gait Trainer Biodex 2, at participant's preferred speed. To eliminate the learning effect, participants practiced at treadmill to determine appropriate gait speed. Once participants implied the preferred speed, they asked to walk at their self selected speed for 6 minutes. Data was recorded between the 2nd and 4th minutes at walk.

SECONDARY OUTCOMES:
Phantom sensation and phantom pain assessment | Initially evaluation at first minute
  Phantom sensation and phantom pain will be asked as existence or not.
Sensory test | Initially evaluation at first minute
  Sensorial loss will be evaluated with Semmes Weinstein Monofilaments (SWME) which is a noninvasive, inexpensive, rapid, and easy-to-apply test and often used in clinical routine assessment. The monofilaments will be applied to the stump along to the incision area and grafted skin area until the monofilaments bended for about one second. Participants will be instructed to say "yes" once they feel the monofilament on their skin. Each test will be repeated for 7 times whether the sensation loss was existed or not. Five true answers from 7 repeat will be accepted as normal feeling. Monofilament tests will beggin at 4.56 as known as protective sensation.